CLINICAL TRIAL: NCT07266844
Title: Evaluating the Safety and Advantages of Using Selective Laser Capsulotomy to Create Capsulorhexis in Cases Intumescent Cataract
Brief Title: CAPSULaser in Cases of Intumescent Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEH-IRB# 432 - 7 - July -2025; Maghrabi eye hospitals (Other: Maghrabi eye hospitals)
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Intumescent Cataract
Keywords: cataract
MeSH Terms: conditions — Cataract | interventions — Posterior Capsulotomy

STUDY DESIGN:
Intervention Model Description: intumescent cataract capsulorhexis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intumescent cataract (Other): CAPSULaser
  Interventions: Procedure: CAPSULaser; Device: capsulotomy

INTERVENTIONS:
Procedure: CAPSULaser — doing capsulotomy using CAPSULaser
Device: capsulotomy — capsulorhexis using CAPSULaser

SUMMARY:
evaluating the use of selective laser in doing capsulotomy in intumescent cataract

DETAILED DESCRIPTION:
Evaluating the safety and advantages of using selective laser capsulotomy for capsulorhexis creation in intumescent cataract

ELIGIBILITY:
Inclusion Criteria:

* patients with intumescent cataract and good pupil dilatation

Exclusion Criteria:

* absence of corneal scaring

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
To measure the actual size compared to result size as measured by slit lamp in mm | 3 months
  To measure the actual size compared to result size as measured by slit lamp
Incidence and number of extended capsulorhexis to the total number of cases | 1 month
  Incidence and number of extended capsulorhexis

CONTACTS AND LOCATIONS:
Locations (1):
- Magrabi eye hospitals, Jeddah, Jedda, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No